CLINICAL TRIAL: NCT01276652
Title: Sleep and Circadian Rhythms in Mechanically Ventilated Patients: a Feasibility and Mechanistic Study.
Brief Title: Sleep and Circadian Rhythms in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); The Brain Research Foundation (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Brian Gehlbach, Clinical Associate Professor of Medicine, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SleepICU111; 5K23HL088020 (NIH)
Record Dates: First submitted 2011-01-10; First posted 2011-01-13 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Failure; Critical Illness
Keywords: Polysomnography; Circadian rhythmicity
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Intervention Model Description: Subjects were randomized in 1:1 fashion to receive the Environmental Modification protocol or usual care. Subsequently a third, observational arm was opened to acquire more physiologic data.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Environmental modification (Active Comparator): Subjects assigned to this group receive the environmental modification intervention for 48 hours beginning the morning after enrollment.
  Interventions: Behavioral: Environmental modification
- Usual care (randomized) (No Intervention): Usual care is provided for the first 48 hours. Subsequently, in the initial protocol, subjects received 48 hours of the environmental modification intervention so long as they remained in the ICU during this time. The opportunity to receive the "Delayed" intervention was later removed from the protocol.
- Usual care (observational) (No Intervention): Usual care was provided.

INTERVENTIONS:
Behavioral: Environmental modification — Environmental modification consists of nursing-related efforts to optimize daytime light exposure, to minimize nighttime light and noise exposure, and to batch nursing care at night.
  Arms: Environmental modification

SUMMARY:
This study examines the feasibility of assessing sleep and circadian rhythmicity in critically ill patients undergoing mechanical ventilation. Secondarily, it will examine the feasibility of reducing subject exposure to environmental light and noise and of delivering routine care according to classical day/night routines.

DETAILED DESCRIPTION:
Over 1 million patients develop respiratory failure annually in the United States; yet, the sleep of patients undergoing mechanical ventilation has received little attention. This protocol enrolls acutely ill medical patients undergoing mechanical ventilation. The feasibility of assessing sleep and circadian rhythmicity through the use of continuous bedside polysomnography and the measurement of core body temperature and urinary hormonal levels at frequent intervals will be explored. As a secondary goal, the feasibility of delivering routine care according to classical day/night routines, and of employing various noise and light reduction strategies at night, will be explored in a subset of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing mechanical ventilation in the medical intensive care unit.

Exclusion Criteria:

* Central nervous system disease (stroke, seizure, dementia, etc)
* Metabolic or hypoxic encephalopathy
* Confirmed or suspected drug overdose
* Currently receiving neuromuscular blockers
* Coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Gehlbach, MD, Principal Investigator — University of Chicago; Jesse Hall, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, there are no plans to share IPD.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the medical ICU at the University of Chicago between November 2001 and December 2008. Subjects were randomized to receive the environmental modification or usual care during the first 48 hours beginning the morning after enrollment. Subsequently, we enrolled 5 subjects in an observational arm (usual care).
Pre-assignment Details: Two subjects were withdrawn by the PI after consent but prior to randomization, when they acutely developed exclusion criteria. One additional subject was withdrawn by the surrogate decision-maker prior to the initiation of the study. No data were collected on these subjects and they are not included in the results.
Groups:
- Randomization: Environmental Modification Group: Subjects randomized to this group underwent the environmental modification intervention designed to promote strong day/night routines for 48 hours.
- Randomization: Usual Care: Subjects received usual care for 48 hours beginning the morning after enrollment. A subset of this group received the intervention on a pilot basis after this time period had elapsed.
- Usual Care (Observational): Subjects received usual care for 48 hours beginning the morning after enrollment.
Period: Period 1: Randomization
Arm/Group | Randomization: Environmental Modification Group | Randomization: Usual Care | Usual Care (Observational)
Started | 9 | 8 | 0 (No subjects were enrolled in this arm during Period 1.)
Completed | 9 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Period 2: Observational
Arm/Group | Randomization: Environmental Modification Group | Randomization: Usual Care | Usual Care (Observational)
Started | 9 | 8 | 5 (Subjects were only enrolled in the Observational arm during Period 2.)
Completed | 9 | 8 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Environmental Modification: Subjects received an environmental modification intervention designed to strengthen day/night routines for the first 48 hours beginning the morning after enrollment. Usual Care was provided outside of this interval. Environmental modification consisted of nursing-related efforts to optimize daytime light exposure, to minimize nighttime light and noise exposure, and to batch nursing care at night.
- Usual Care (Randomized); Usual Care (Observational): Usual Care was provided for the first 48 hours.
- Total: Total of all reporting groups
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational) | Total
Number analyzed (Participants) | 9 | 8 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (22.7) | 59.4 (16.8) | 65.8 (6.0) | 62.2 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 4 | 3 | 2 | 9
APACHE II score [Mean (Standard Deviation); unit: units on a scale] — The Acute Physiology and Chronic Health Evaluation II score is designed to measure the severity of illness of patients admitted to intensive care units, with higher scores indicating patients who are more likely to die during the admission. The score is an integer score that ranges from 0 to 71 and is calculated within 24 hours of admission from the patient's age, routinely collected physiologic data, and information regarding the patient's chronic health status.
  units on a scale | 22.7 (6.6) | 21.0 (8.0) | 19.2 (6.5) | 20.9 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Successfully Undergo Continuous Bedside Polysomnography for at Least 24 Hours.
Description: This study assesses the feasibility of studying sleep and circadian rhythmicity in acutely ill, mechanically ventilated patients through the application of continuous bedside polysomnography. Feasibility will be assessed by determining the percentage of enrolled subjects who undergo at least 24 hours of continuous bedside polysomnography.
Time Frame: Average 4 days (patients followed to hospital discharge)
Measure: Count of Participants; unit: Participants
Groups:
- Environmental Modification: A subset of subjects were randomly assigned to receive an environmental modification intervention either early (first 48 hrs) or late (next 48 hrs). Usual Care was provided outside of this interval. Environmental modification consisted of nursing-related efforts to optimize daytime light exposure, to minimize nighttime light and noise exposure, and to batch nursing care at night.
- Usual Care (Randomized): Usual Care was provided during the first 48 hours.
- Usual Care (Observational): Usual care was provided for 48 hours.
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
Number analyzed (Participants) | 9 | 8 | 5
Participants | 9 | 8 | 5

2. Secondary Outcome: Subject Tolerance of the Environmental Modification Protocol
Description: This outcome measure will examine, in a preliminary fashion, subject tolerance of the environmental modification protocol. Tolerance will be assessed through qualitative interviews performed by the PI with the subjects.
Time Frame: Average 4 days (patients followed to hospital discharge)
Population: Only subjects who received the intervention were assessed.
Measure: Number; unit: Subjects who tolerated the protocol
Groups:
- Environmental Modification: In a subset of this study, subjects are randomly assigned to receive an environmental modification intervention either early (first 48 hrs) or late (next 48 hrs). Usual Care was provided outside of this interval.
  Environmental modification: Environmental modification consists of nursing-related efforts to optimize daytime light exposure, to minimize nighttime light and noise exposure, and to batch nursing care at night.
- Usual Care (Randomized): Usual care for 48 hours.
- Usual Care (Observational): Usual care is provided to the subjects for 48 hours.
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
Number analyzed (Participants) | 9 | 0 | 0
Subjects who tolerated the protocol | 9 |  |

3. Other Pre Specified Outcome: Occurrence of REM Sleep
Description: Occurrence of identifiable rapid eye movement (REM) sleep in each subject.
Time Frame: Average 4 days (patients followed to hospital discharge)
Population: In one subject in the environmental modification group, the files were lost after acquisition and this analysis was unable to be performed.
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care (Randomized); Usual Care (Observational): Usual Care was provided to the subjects.
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
Number analyzed (Participants) | 8 | 8 | 5
Participants | 2 | 0 | 0

4. Other Pre Specified Outcome: Normal Timing of 6-sulfatoxymelatonin Excretion
Description: The number of participants in each group who exhibit normal timing of 6-sulfatoxymelatonin excretion will be reported. The normal timing of peak melatonin excretion was considered to be between midnight and 05:00. Subjects in whom the melatonin onset occurred after midnight or the acrophase occurred after 05:00 were considered to be phase delayed, while patients whose acrophase occurred prior to midnight were considered to be phase advanced.
Time Frame: Average 4 days (patients followed to hospital discharge)
Population: 24-hour 6-sulfatoxymelatonin profiles were successfully collected in 16 subjects total. In one subject in the usual care (observational) group, there were insufficient data to determine melatonin timing.
Measure: Count of Participants; unit: Participants
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
Number analyzed (Participants) | 5 | 6 | 4
Participants | 1 | 2 | 1

5. Post Hoc Outcome: Presence of Normal Slow Wave Activity
Description: Slow wave activity in health exhibits diurnal and ultradian periodicity and a homeostatic decline at night. The number of subjects exhibiting these characteristics was calculated for each group.
Time Frame: Average 4 days (patients followed to hospital discharge)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
Number analyzed (Participants) | 8 | 8 | 5
Participants | 0 | 0 | 0

6. Post Hoc Outcome: Presence of Normal Spectral Edge Frequency 95% (SEF95) Activity
Description: SEF95 is normally higher during wakefulness during sleep. The normal sleep SEF95 profile is rhythmic with an approximately 90 minute periodicity. We analyzed the number of subjects who exhibited this normal profile.
Time Frame: Average 4 days (patients followed to hospital discharge)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
Number analyzed (Participants) | 8 | 8 | 5
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Until ICU discharge, an average of 1 week.
Groups:
- Environmental Modification: Environmental modification is provided for the initial 48 hours and consists of nursing-related efforts to optimize daytime light exposure, to minimize nighttime light and noise exposure, and to batch nursing care at night.
- Usual Care (Randomized); Usual Care (Observational): Usual care is provided to the subjects.
Arm/Group | Environmental Modification | Usual Care (Randomized) | Usual Care (Observational)
All-Cause Mortality (participants affected / at risk) | 2/9 | 2/8 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/5

LIMITATIONS AND CAVEATS:
Logistical issues related to the performance of continuous bedside polysomnography may vary from institution to institution, thereby limiting the generalizability of our results where the primary outcome measure is concerned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No